CLINICAL TRIAL: NCT03431233
Title: An Exploratory Study of the Effect of Premeal Consumption of Protein-enriched, Dietary Fiber-fortified Cereal Bar on Food Intake in Healthy Subjects
Brief Title: Effect of Premeal Protein-bar on Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Young Min Cho, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H-1705-091-855
Record Dates: First submitted 2018-01-15; First posted 2018-02-13 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Healthy Subjects
Keywords: protein-enriched bar; food intake; appetite; satiety related hormones
MeSH Terms: interventions — Water

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1 (Experimental): protein enriched bar->commercial cereal bar->water
  Interventions: Dietary Supplement: Protein-enriched bar, commercial cereal bar, or water
- Group 2 (Experimental): protein enriched bar->water->commercial cereal bar
  Interventions: Dietary Supplement: Protein-enriched bar, commercial cereal bar, or water
- Group 3 (Experimental): commercial cereal bar->protein enriched bar->water
  Interventions: Dietary Supplement: Protein-enriched bar, commercial cereal bar, or water
- Group 4 (Experimental): commercial cereal bar->water->protein enriched bar
  Interventions: Dietary Supplement: Protein-enriched bar, commercial cereal bar, or water
- Group 5 (Experimental): water->protein enriched bar->commercial cereal bar
  Interventions: Dietary Supplement: Protein-enriched bar, commercial cereal bar, or water
- Group 6 (Experimental): water->commercial cereal bar->protein enriched bar
  Interventions: Dietary Supplement: Protein-enriched bar, commercial cereal bar, or water

INTERVENTIONS:
Dietary Supplement: Protein-enriched bar, commercial cereal bar, or water — Protein enriched bar, commercial cereal bar, or water will be provided 15 minutes before breakfast.

SUMMARY:
The aim of this study is to explore premeal protein-enriched bar effect in food intake in healthy subjects.

DETAILED DESCRIPTION:
Twenty healthy subjects will be recruited. Every subject will be randomized in 6 groups and studied on 3 separate days in random order with 1 week intervals. These participants will consume protein enriched bar, commercial cereal bar, or water followed by a standardized diet (gimbap). For study outcomes, food intake, appetite and satiety (visual analog scale), plasma glucose, and satiety related hormone will be measured. Blood sampling will be done before 15 min of breakeast, at the moment of start of breakfast (0 min), and then 30, 60, 90, 120 min. Plasma glucose levels, total/active GLP-1, ghrelin, total PYY will be measured.

ELIGIBILITY:
* Inclusion Criteria:

  * BMI 18.5~35 kg/m2
  * Never diagnosed by diabetes
  * Fasting plasma glucose <=100mg/dl and HbA1c <6.0%
* Exclusion Criteria:

  * Those who diagnosed by Type 1 or Type 2 diabetes
  * Allergy to wheat, flour, nuts, milk
  * Pregnancy/lactation
  * AST or ALT >2.5 times of upper normal reference range
  * eGFR <30 mL/min/1.73m2
  * Hb <10g/dl
  * History of GI surgery (except hemorrhoidectomy, appendectomy)

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Food intake | 120min
  grams and caloric intake of standardized gimbap

SECONDARY OUTCOMES:
Appetite (visual analogue scale : score 1 to 10) | 120min
  (1: I am not hungry at all, 10: I have never been more hungry)
Satiety (visual analogue scale : score 1 to 10) | 120min
plasma glucose (mmol/L) | -15min, 0(breakfast), 30, 60, 90, 120 min
  plasma level of glucose
plasma active/total GLP-1 (pmol/L) | -15min, 0(breakfast), 30, 60, 90, 120 min
  plasma level of active/total GLP-1
plasma active ghrelin (ng/ml) | -15min, 0(breakfast), 30, 60, 90, 120 min
  plasma level of active ghrelin
plasma total peptide YY (pg/ml) | -15min, 0(breakfast), 30, 60, 90, 120 min
  plasma level of peptide YY

CONTACTS AND LOCATIONS:
Overall Officials: Young Min Cho, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea